CLINICAL TRIAL: NCT00255775
Title: Evaluation of the Biological Effects of Broccoli Sprout Extract in Smokers
Brief Title: Broccoli Sprout Extract in Preventing Lung Cancer in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Prevention
Other Study IDs: JHOC-J0427, CDR0000450158; P50CA058184 (NIH); P30CA006973 (NIH); JHOC-J0427; JHOC-04051801; NCT00090350 (obsolete NCT alias)
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2010-08

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

INTERVENTIONS:
Dietary Supplement: broccoli sprout extract
Procedure: complementary or alternative medicine procedure

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs or substances to keep cancer from forming, growing, or coming back. The use of broccoli sprout extract may prevent lung cancer.

PURPOSE: This clinical trial is studying how well broccoli sprout extract works in preventing lung cancer in smokers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the effect of broccoli sprout extract on levels of DNA adducts in participants who smoke.
* Determine the effectiveness of broccoli sprout extract in reducing tobacco-carcinogen induced DNA adducts in these participants.

Secondary

* Determine the effects of broccoli sprout extract on markers of the Nrf2 pathway in these participants.
* Determine the effectiveness of broccoli sprout extract, in increasing the activity of the Nrf2 pathway, in these participants.
* Evaluate the feasibility of using lymphocytes and buccal cells to monitor DNA adducts and changes in the Nrf2 pathway in these participants.

OUTLINE: Participants are stratified according to GST genotypic polymorphism (M1 vs T1).

Participants receive oral broccoli sprout extract daily for 3 weeks. Participants keep a daily diary of their eating and smoking habits for 3 weeks before, during, and for 3 weeks after study treatment. They must continue to smoke during the study, but are encouraged to quit after completing the study treatment.

PROJECTED ACCRUAL: A total of 70 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current smoker with ≥ 30 pack-year history of smoking

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 4,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile participants must use effective contraception
* No other medical condition that would preclude study treatment or compliance
* No gastrointestinal condition that would affect absorption, preclude taking oral medication, or necessitate IV alimentation

PRIOR CONCURRENT THERAPY:

Surgery

* No prior surgery affecting absorption

Other

* More than 6 weeks since prior vitamins, herbal supplements, non-steroidal anti-inflammatory drugs, or antibiotics
* No concurrent dietary intake of cruciferous vegetables

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States